CLINICAL TRIAL: NCT02280629
Title: Randomized, Double-blind, Double-dummy, Placebo-controlled, Phase III Clinical Trial on the Efficacy and Safety of a 48-weeks Treatment With Gastro-resistant Phosphatidylcholine (LT-02) Versus Placebo Versus Mesalamine for Maintenance of Remission in Patients With Ulcerative Colitis
Brief Title: Phosphatidylcholine (LT-02) vs. Placebo vs. Mesalamine for Maintenance of Remission in Ulcerative Colitis (PROTECT-2)
Acronym: PROTECT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCG-4/UCR; 2013-001205-84 (EudraCT Number)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LT-02 (Experimental): LT-02 1.6g twice daily AND mesalamine PLACEBO three-times daily
  Interventions: Drug: LT-02
- Placebo (Placebo Comparator): LT-02 PLACEBO twice daily AND mesalamine PLACEBO three-times daily
  Interventions: Drug: Placebo
- Mesalamine (Active Comparator): LT-02 PLACEBO twice daily AND 500mg mesalamine PLACEBO three-times daily
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: LT-02 — LT-02 1.6g twice daily AND mesalamine PLACEBO three-times daily
  Arms: LT-02
Drug: Placebo — LT-02 PLACEBO twice daily AND mesalamine PLACEBO three-times daily
  Arms: Placebo
Drug: Mesalamine — LT-02 PLACEBO twice daily AND mesalamine 500mg three-times daily
  Arms: Mesalamine

SUMMARY:
The purpose of this study is to prove the superiority of a 48-weeks treatment with 3.2 g/day delayed-release phosphatidylcholine (LT-02) versus placebo for the maintenance of remission in patients with ulcerative colitis (UC)

ELIGIBILITY:
Major Inclusion Criteria:

* Signed informed consent
* Men or women, 18 to 70 years of age
* Historically confirmed diagnosis of UC by endoscopy and histology
* Patients being in clinical and endoscopical remission at baseline
* Negative pregnancy test in females of childbearing potential at baseline visit

Major Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ischemic colitis, radiation colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis), diverticular disease associated colitis
* Toxic megacolon or fulminant colitis
* Colon resection
* Malabsorption syndromes
* Celiac disease
* Bleeding hemorrhoids
* Other inflammatory or bleeding disorders of the colon and intestine, or diseases that may cause diarrhea or gastrointestinal bleeding
* History or presence of ischemic heart disease, myocardial infarction, peripheral arterial disease, ischemic stroke, or transient ischemic attack
* Any severe concomitant renal, endocrine, or psychiatric disorder, which in the opinion of the investigator might have an influence on the patient's compliance or the interpretation of the results
* Any relevant known systemic disease (e.g., AIDS, active tuberculosis)
* Severe co-morbidity substantially reducing life expectancy
* History of cancer in the last five years
* Abnormal hepatic function at screening visit, liver cirrhosis
* Abnormal renal function at screening visit
* Patients with known hypersensitivity to soy
* Known intolerance/hypersensitivity to Investigational Medicinal Product (IMP: LT-02 or mesalamine)
* Treatment with steroids (oral, inhalative, or intravenous [IV]), cyclosporine or tacrolimus within last 4 weeks prior to randomization
* Treatment with methotrexate within last 6 weeks prior to randomization
* Treatment with TNF-alpha-antagonists, azathioprine, 6-mercaptopurine, or anti-integrin therapy within last 8 weeks prior to randomization
* Treatment with rectal mesalamine or corticosteroid formulations within last 2 weeks prior to randomization
* Treatment with other investigational drug within last 12 weeks prior to randomization except LT-02
* Existing or intended pregnancy or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who are relapse-free and are not a treatment failure | 48 weeks

SECONDARY OUTCOMES:
Mean change from baseline in the total mDAI | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Dignass, Prof Dr, Principal Investigator — Agaplesion Markus Krankenhaus
Locations (1):
- Agaplesion Markus-Krankenhaus, Frankfurt a.M., Germany

REFERENCES:
- [Derived] Dignass A, Stremmel W, Horynski M, Poyda O, Armerding P, Fellermann K, Langhorst J, Kuehbacher T, Uebel P, Stein J, Novacek G, Avalueva E, Oliinyk O, Hasselblatt P, Dorofeyev A, Heinemann H, Mueller R, Greinwald R, Reinisch W; International PROTECT-1/2 Study Groups. Modified-Release Phosphatidylcholine (LT-02) for Ulcerative Colitis: Two Double-Blind, Randomized, Placebo-Controlled Trials. Clin Gastroenterol Hepatol. 2024 Apr;22(4):810-820.e7. doi: 10.1016/j.cgh.2023.09.031. Epub 2023 Oct 6. PMID 37806372